CLINICAL TRIAL: NCT06913803
Title: To Find Effectiveness of Stretching Versus Soft Tissue Mobilization in Coccydynia in Postpartum Females
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/809
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Coccidioidomycosis
MeSH Terms: conditions — Coccidioidomycosis | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching (Experimental)
  Interventions: Diagnostic Test: Stretching
- Soft Tissue Mobilization (Experimental)
  Interventions: Combination Product: Soft Tissue Mobilization

INTERVENTIONS:
Diagnostic Test: Stretching — The group A contains 34 patients and received STM for twice a week for three weeks with each session lasting approximately 20 min.focusing on mobilizing soft tissue to enhance circulation, reduce scar tissue and improve tissue flexibility.
  Arms: Stretching
Combination Product: Soft Tissue Mobilization — Group B received both STM and stretching twice a week for three weeks with each session lasting approximately 20 min.encourage the patient to breathe deeply and slowly to promote relaxation.The stretching of tight muscles 1 set of 10 repetitions hold of 5 second of each exercise,then breathing for 1 min
  Arms: Soft Tissue Mobilization

SUMMARY:
This research is to determine the effectiveness of stretching versus soft tissue mobilization in coccydynia patients.The main purpose of the study is the the development of evidence based therapeutic protocols for postpartum coccydynia patients to improve functional impairment, range of motion, and reduction of pain.

DETAILED DESCRIPTION:
The study design is randomized controlled trial.The interventions were carried out twice a week for three weeks with each session lasting approximately 20 min.Group A contains 34 patients and received STM focusing on mobilizing soft tissue to enhance circulation reduce scar tissue and improve functional flexibility.Group B received both STM and stretching twice a week for three weeks with each session lasting approximately 20 min.During entire treatment the therapist kept close eye on patient discomfort.The significance of the study lies in it's potential to enhance more effective non invasive treatment to alleviate symptoms

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by orthopedic surgeon with sign and symptoms of coccydynia and radiograph X ray for confirmation.: postpartum females after 2 to 3 months after delivery
* office working females
* aged 20 to 35 years
* females with c section

Exclusion Criteria:

* FEMALES with vaginal delivery
* experience severe post operative pain
* active pelvic or abdominal infections
* ovarian cyst, fibroids,or obstructive endometrial polyps
* neurological conditions

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE(NPRS) | 12 Months
  The Numeric Pain Rating Scale (NPRS) is a widely used, 11-point scale (0-10) for measuring pain intensity, with 0 representing "no pain" and 10 representing "worst pain imaginable
Oswestry Disability Index (ODI) | 12 Months
  The Oswestry Disability Index (ODI) scores disability levels related to low back pain on a scale of 0 to 100, with 0 indicating no disability and 100 representing the highest level of disability

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Ganga Ram Hospital Physiotherapy department , Mozang, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No